CLINICAL TRIAL: NCT05195710
Title: Preoperative Y-90 Radioembolization for Tumor Control and Future Liver Remnant Hypertrophy in Patients With Colorectal Liver Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0521; NCI-2021-13239 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-11-24; First posted 2022-01-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yttrium-90 (Experimental): Help to control the tumor(s) on the right side of the liver while the remaining left side of the liver, which is clear of cancer, grows.
  Interventions: Drug: Yttrium-90 (Y-90) resin microspheres

INTERVENTIONS:
Drug: Yttrium-90 (Y-90) resin microspheres — Given by scan

SUMMARY:
A prospective, interventional study evaluating the safety of Y-90 TARE for tumor control of the right side and induction of left liver hypertrophy as part of a planned single-stage or two-stage hepatectomy for patients with CLM and insufficient FLR at the time of presentation.

DETAILED DESCRIPTION:
Primary Objective:

To examine the safety and feasibility of Y-90 TARE directed to the right hemi-liver for induction of left liver FLR hypertrophy as part of a planned hepatectomy for patients with CLM.

Secondary Objectives:

* To describe changes in liver volume after Y-90 TARE, including:

  * The kinetic growth rate (KGR) of the FLR
  * Degree of hypertrophy 6 weeks after TARE
  * Atrophy of targeted right hemi-liver from TARE date to date of surgery
* To describe additional interventional procedures needed to induce additional hypertrophy if insufficient hypertrophy from Y-90 TARE
* To assess the proportion of TARE patients who undergo attempted and complete curative-intent resection of CLM
* To assess measures of disease control, including:

  * Tumor marker trend
  * RECIST/mRECIST criteria
  * CT morphologic response
  * PET CT response
* To describe Patient Reported Outcomes using MDASI-GI
* To assess FLR liver quality, right-sided surgical adhesions from TARE intraoperatively
* To describe dosimetry of individual liver lesions - using SPECT/CT, CT, and pathology correlation
* To describe change in liver function measured by the pre- and post-TARE HIDA SPECT/CT scans and hepatic function blood tests

ELIGIBILITY:
Inclusion Criteria:

* Borderline resectable unresectable (due to insufficient liver volume at presentation) colorectal liver metastases with potential curative intent, as determined by the surgeon and multidisciplinary team
* Anticipated standardized FLR (sFLR) that would require right portal vein embolization (PVE) to increase the sFLR prior to either a single major hepatectomy, or prior to the second stage hepatectomy as part of a two-stage hepatectomy strategy, all in the setting of curative-intent resection(s). This evaluation will be documented in the clinical chart
* Received at least four cycles (or two months) of chemotherapy
* Willing, able and mentally competent to provide written informed consent
* Medically and physically operable as determined by the surgeon

Exclusion Criteria:

* Extrahepatic disease that precludes intended curative intent treatment sequencing (treatable primary tumor and lung metastases allowed). "Treatable" is defined as having an intended future plan for local therapy (surgery, radiation, or ablation) as determined by the patient's medical oncologist and surgical oncologist
* Projected sFLR before Y-90 of <20% (starting with sFLR that is unrealistic for improvement to ≥30%)
* Performance status limitations (Karnofsky <80%, ECOG >1)
* Portal hypertension and/or cirrhosis
* Starting total bilirubin >1.3 mg/dL (except if patient has Gilbert's Disease)
* CEA >200 after 4 cycles of chemotherapy upon restaging visit
* Clinical progression of disease on imaging and/or tumor marker after 4 cycles of chemotherapy that is clinically judged by surgical oncology and medical oncology to preclude surgical resection
* Platelet count <100,000/µL
* Albumin <3.5 g/dl
* Symptomatic primary colon or rectal cancer (without pre-existing proximal diverting ostomy)
* Pregnant or breast-feeding patient
* Other medical or clinical contraindications to liver surgery
* Non-English-speaking participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The evaluation from using the feasibility of Y-90 TARE directed to the right hemi-liver for induction of left liver FLR hypertrophy as part of a planned hepatectomy for patients with CLM. | through study completion, an average of 1 year
The evaluation of using the safety of Y-90 TARE directed to the right hemi-liver for induction of left liver FLR hypertrophy as part of a planned hepatectomy for patients with CLM. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Wei Tzeng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org